CLINICAL TRIAL: NCT07164391
Title: Empowering Vietnamese Americans: A Culture-Centric Digital Storytelling Intervention to Boost HPV Vaccination
Brief Title: Empowering Vietnamese Americans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Angela Chia-Chen Chen, Professor & Endowed Chair, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IP00769244
Record Dates: First submitted 2025-06-09; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HPV Vaccination; Cancer Prevention
Keywords: HPV; cancer prevention; Vietnamese American; youth; digital storytelling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Story group (Active Comparator): This group will receive the digital Intervention for Vietnamese-American Storytelling (VIDAS)
  Interventions: Behavioral: Digital Intervention for Vietnamese-American Storytelling (VIDAS)
- Video group (Active Comparator): This group will receive the HPV Educational Video Intervention.
  Interventions: Behavioral: HPV Educational Video Intervention
- Teen General Health group (Placebo Comparator): This group will receive the Teen General Health intervention.
  Interventions: Behavioral: Teen General Health

INTERVENTIONS:
Behavioral: Digital Intervention for Vietnamese-American Storytelling (VIDAS) — The intervention consists of 4 brief stories about HPV vaccine, created by Vietnamese mothers
  Arms: Story group
Behavioral: HPV Educational Video Intervention — The intervention consists of 4 brief informational videos about HPV and the vaccine
  Arms: Video group
Behavioral: Teen General Health — This intervention consists of 4 brief videos on general teen health topics, such as mental health, social media usage.
  Arms: Teen General Health group

SUMMARY:
The goal of this clinical trial is to learn whether short videos can help Vietnamese American mothers decide to vaccinate their children against HPV (human papillomavirus). The study will explore: (1) which type of video is most effective in encouraging mothers to vaccinate their children; (2) how mothers perceive and engage with the videos; and (3) how many children receive the HPV vaccine after their mothers watch the videos.

Participants will be randomly assigned to one of three groups: (a) watch four short digital stories about the HPV vaccine created by Vietnamese mothers; (b) watch four short informational videos about HPV and the vaccine; or (c) watch four short videos on general teen health topics such as mental health and social media use. Participants will complete brief surveys and their child's HPV vaccination status will be checked two months after the intervention.

DETAILED DESCRIPTION:
This study focuses on increasing HPV vaccination rates among Vietnamese American (VA) youth by engaging their mothers-who are key decision-makers-in culturally relevant video interventions. VA females experience disproportionately high rates of HPV-related cervical cancer and low vaccine uptake. Contributing factors include limited HPV knowledge, low English proficiency, and culturally influenced health beliefs. There is a critical need for tailored, community-driven interventions to address these disparities.

Researchers will evaluate three different 4-week video-based interventions: a digital storytelling (DST) intervention featuring personal stories created by Vietnamese mothers, an informational HPV video series, and a general teen health video series. Each mother will view one 3-minute video per week over four weeks. The study uses a randomized, 3-arm design with 60 VA mothers of unvaccinated children ages 11-14 assigned to one of the three groups.

The study draws on the Theory of Planned Behavior and a culture-centric health promotion framework. It aims to measure feasibility, acceptability, and changes in vaccination intention and behavior. Follow-up assessments will occur two months post-intervention to evaluate vaccine uptake. Additionally, a subset of participants will complete interviews to explore engagement and refine future trial design.

Data will be collected at baseline, post-intervention, and 2-month follow-up using online surveys and secure platforms. To ensure equitable participation, the study incorporates bilingual staff, culturally tailored outreach, community partnerships, and graduated incentives. Findings will inform future large-scale trials and may help scale culturally grounded HPV prevention strategies for other underserved populations.

ELIGIBILITY:
Inclusion Criteria: An individual is eligible if they:

* Self-identify as a Vietnamese American or immigrant woman aged 18 years or older
* Are the primary caregiver of at least one unvaccinated child aged 11-14 years
* Can speak and read English
* Agree to receive text messages and/or emails related to project activities during the study period

Exclusion Criteria:

* inability/unwillingness to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Child's HPV vaccine initiation | 2-month follow up (T2)
  Whether the target child receives the 1st HPV vaccine
Mother's intention to vaccinate the eligible child against HPV | T0 (baseline), T1 (immediately post intervention), T2 (2-month follow up)
  One item to measure mother's intention to vaccinate the eligible child against HPV

IPD SHARING:
Plan to Share IPD: Undecided
Privacy and ethical issues